CLINICAL TRIAL: NCT06641830
Title: A Pediatric Cardiomyopathy Cohort Study: the Emerging Role of CMR in Clinical Practice
Brief Title: A Integrated Study in Pediatric Patients with Cardiomyopathy
Status: Enrolling by invitation | Type: Observational
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Ling-Yi Wen, Principal Investigator, West China Second University Hospital
Other Study IDs: WestChinaSUH2024222
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Pediatric Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The whole boold including blood cell and plasma will be collected for laboratory and genetic test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- pediatric patients with cardiomyopathy

SUMMARY:
This observational study aims to manage children with cardiomyopathy in the long term. It collects baseline data, laboratory test data, and medical imaging data during the hospitalization and follow-up.

During their disease progress, participants will undergo cardiovascular magnetic resonance, echocardiography, electrocardiography, laboratory tests, and when hospitalization and follow-up, and the baseline data will be collected in the admission. All the above examination data will be analysed to assess the clinical characteristics, current status of diagnosis and treatment, and the prognostic risk factors for children with cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients diagnosed with cardiomyopathy.

Exclusion Criteria:

* a history of cardiovascular disease ( such as congenital heart disease, cardiomyopathy, rheumatic heart disease, valvular disease ).
* Mentally abnormal.
* Poor compliance.
* Heart, kidney and other important organs were seriously incomplete.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: From the past to Jaunary 2034, pediatric patients diagnosed with cardiomyopathy were recruited from West China Second University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2034-01-01 (Estimated); Study Completion 2034-09-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 10 years after the onset
  Major adverse cardiovascular events including cardiac death, transient ischemic attack or stroke, myocardial infarction, arrhythmia, heart failure, severe valvular disease, percutaneous coronary intervention, coronary artery bypass graft, and other cardiovascular surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mazzarotto F, Hawley MH, Beltrami M, Beekman L, de Marvao A, McGurk KA, Statton B, Boschi B, Girolami F, Roberts AM, Lodder EM, Allouba M, Romeih S, Aguib Y, Baksi AJ, Pantazis A, Prasad SK, Cerbai E, Yacoub MH, O'Regan DP, Cook SA, Ware JS, Funke B, Olivotto I, Bezzina CR, Barton PJR, Walsh R. Systematic large-scale assessment of the genetic architecture of left ventricular noncompaction reveals diverse etiologies. Genet Med. 2021 May;23(5):856-864. doi: 10.1038/s41436-020-01049-x. Epub 2021 Jan 26. PMID 33500567
- [Background] Bogle C, Colan SD, Miyamoto SD, Choudhry S, Baez-Hernandez N, Brickler MM, Feingold B, Lal AK, Lee TM, Canter CE, Lipshultz SE; American Heart Association Young Hearts Pediatric Heart Failure and Transplantation Committee of the Council on Lifelong Congenital Heart Disease and Heart Health in the Young (Young Hearts). Treatment Strategies for Cardiomyopathy in Children: A Scientific Statement From the American Heart Association. Circulation. 2023 Jul 11;148(2):174-195. doi: 10.1161/CIR.0000000000001151. Epub 2023 Jun 8. PMID 37288568
- [Background] Arbelo E, Protonotarios A, Gimeno JR, Arbustini E, Barriales-Villa R, Basso C, Bezzina CR, Biagini E, Blom NA, de Boer RA, De Winter T, Elliott PM, Flather M, Garcia-Pavia P, Haugaa KH, Ingles J, Jurcut RO, Klaassen S, Limongelli G, Loeys B, Mogensen J, Olivotto I, Pantazis A, Sharma S, Van Tintelen JP, Ware JS, Kaski JP; ESC Scientific Document Group. 2023 ESC Guidelines for the management of cardiomyopathies. Eur Heart J. 2023 Oct 1;44(37):3503-3626. doi: 10.1093/eurheartj/ehad194. No abstract available. PMID 37622657
- [Background] Lipshultz SE, Law YM, Asante-Korang A, Austin ED, Dipchand AI, Everitt MD, Hsu DT, Lin KY, Price JF, Wilkinson JD, Colan SD. Cardiomyopathy in Children: Classification and Diagnosis: A Scientific Statement From the American Heart Association. Circulation. 2019 Jul 2;140(1):e9-e68. doi: 10.1161/CIR.0000000000000682. Epub 2019 May 28. PMID 31132865
- [Background] Lee TM, Hsu DT, Kantor P, Towbin JA, Ware SM, Colan SD, Chung WK, Jefferies JL, Rossano JW, Castleberry CD, Addonizio LJ, Lal AK, Lamour JM, Miller EM, Thrush PT, Czachor JD, Razoky H, Hill A, Lipshultz SE. Pediatric Cardiomyopathies. Circ Res. 2017 Sep 15;121(7):855-873. doi: 10.1161/CIRCRESAHA.116.309386. PMID 28912187